CLINICAL TRIAL: NCT03887494
Title: Prospective Multi-center Study of Impact of Femoral "Y-strut" Implant on Pain and Quality of Life in Patients With Lytic Bone Metastases of the Femoral Neck
Brief Title: Study of the Impact of the Femoral Implant "Y-strut" on Lytic Bone Metastases of the Femoral Neck (WAZA-ARY)
Acronym: WAZA-ARY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hyprevention (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K171014J; 2018-A01901-54 (Other: Eudract Number)
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Neoplasms, Bone Tissue; Pain, Intractable; Hip Fractures
Keywords: Implantable device, Hip fractures
MeSH Terms: conditions — Neoplasms, Bone Tissue; Pain, Intractable; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Y-Strut Implant (Experimental): Single interventional arm
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — Implantation of Y-Strut + cementoplasty in the femoral neck

SUMMARY:
Bone metastases appear in many cancers. They are associated with severe pain that is refractory to standard treatment. Improving the quality of life and better pain relief is therefore an essential goal of the treatment of metastatic disease. The most common site of long bone metastases is the superior femoral epiphysis.

The usual management of patients with bone metastases in the superior femoral epiphysis is based on gamma implant osteosynthesis when there is a known risk of fracture (Mirels score> 8). Nonetheless this surgery is only accessible to a few patients because of the associated morbidities.

Percutaneous cementoplasty has been developed to treat patients who are not eligible for conventional surgery. It consists in a filling of the bone cavity created by metastasis using an acrylic resin. However, these approaches do not completely prevent the risk of upper femoral epiphyseal fracture due to the low mechanical resistance of the resin to shear movements.

The Y-STRUT® implantable medical device was developed to overcome this risk of superior femoral epiphyseal fracture by the biomechanical strengthening of the proximal femur in addition to cementoplasty. It has been successfully tested in more than 70 patients with cancer but access to reimbursement and the APHP market have been postponed due to lack of sufficient clinical evidence.

The investigators propose this prospective phase 2a study in order to provide evidence of the performance of the Y-STRUT® implant.

DETAILED DESCRIPTION:
The design consists in a multicenter national open simple arm trial.

All eligible patients with a lytic bone metastases of the superior femoral epiphysis will be included.

The main objective of this study is to describe the impact of the Y-STRUT® implant on the quality of life of patients with lytic bone metastases of the femoral neck by comparing quality of life scores before and one month after the intervention of implantation of the implant.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* patient with a lytic or mixed matrix bone metastasis of the superior femoral epiphysis visualized in imaging
* MIRELS score ≥8 within 20 days prior to inclusion,
* ECOG-PS 2 or 3 within 20 days prior to inclusion,
* Cervico-diaphyseal angle between 115 ° and 135 ° inclusive,
* Length of the proximal part of the femur greater than or equal to 90 mm
* Patient refusing gamma nail
* Life expectancy greater than 6 months

Exclusion Criteria:

* Act of general anesthesia impossible,
* ECOG <2 (patients eligible for nailing treatment),
* INR <0.7 in the 24 hours preceding the intervention,
* Platelets <70000 / mm3 within 24 hours of surgery,
* Allergy previously known by the patient to PEEK and / or PMMA,
* Patient who previously had a cementoplasty of the target lesion,
* Osteolysis of the target epiphyseal cortex> 2/3 of the circumference of the epiphyseal cortex,
* Pre-fracture lesions of the underlying ipsilateral diaphysis or ipsilateral acetabulum
* Patient unable or unwilling to give written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-09-06 (Estimated); Primary Completion 2020-05-22 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure of Quality of Life for each patient within one month after the implantation | 30 days
  Measure of the Quality of Life score using the questionary of quality of life of the European Organization for Research and Treatment of Cancer BM-22.
  Patients answer at 22 questions to describe their quality of life during the past week. For each question, patient must choose between 1.not at all, 2.a little, 3.enough, 4.a lot. A global score is calculated by adding the 22 score of each questions. The higher value of this global score represents the better outcome.

SECONDARY OUTCOMES:
Target lesion fracture within one month after the implantation | 30 days
  Number of target lesion fracture
Target lesion fracture within 2 months after the implantation | 2 months
  Number of target lesion fracture
Non-target femoral fracture within 2 months after the implantation | 2 months
  Number of Non-target femoral fracture
Non-target femoral fracture within one month after the implantation | 30 days
  Number of Non-target femoral fracture
Analgesic medication needs (type and dose) within one month after the implantation | 30 days
  Consumption of analgesic medication
Analgesic medication needs (type and dose) within 2 months after the implantation | 2 months
  Consumption of analgesic medication
total AE/SAE within one month after the implantation | 30 days
  Number of AE/SAE
total AE/SAE within 2 months after the implantation | 2 months
  Number of AE/SAE
AE/SAE imputable to the device (number) within one month after the implantation | 30 days
  Number of AE/SAE imputable to the device
AE/SAE imputable to the device (number) within 2 months after the implantation | 2 months
  Number of AE/SAE imputable to the device
AE/SAE imputable to the implatation (number) within one month after the implantation | 30 days
  Number of AE/SAE imputable to the implatation
AE/SAE imputable to the implatation (number) within 2 months after the implantation | 2 months
  Number of AE/SAE imputable to the implatation
Morphinic mean dose per day within one month after the implantation | 30 days
  Consumption of morphinic mean dose per day during the month after the procedure
Morphinic mean dose per day within 2 months after the implantation | 2 months
  Consumption of morphinic mean dose per day during the 2 months after the procedure
Quality of Life score (EORTC QLQ BM-22) within 2 months after the implantation | 2 months
  Measure of the Quality of Life score using the questionary of quality of life of the European Organization for Research and Treatment of Cancer BM-22.
  Patients answer at 22 questions to describe their quality of life during the past week. For each question, patient must choose between 1.not at all, 2.a little, 3.enough, 4.a lot. A global score is calculated by adding the 22 score of each questions. The higher value of this global score represents the better outcome.
Pain score at target site within 2 months after the implantation: VAS | 2 months
  Use of Visual Analog Scale (VAS) to evaluate the pain at target site (between 0: no pain to 10: intolerable pain)
Length of stay within 2 months after the implantation | 2 months
  Length of stay at hospital
Exit mode of hospital within 2 months after the implantation | 2 months
  at home, re-education unit

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Pellerin, MD, PhD, Principal Investigator — AP-HP, Hôpital Européen Georges Pompidou, Paris; François Cornelis, MD, PhD, Principal Investigator — AP-HP, Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying published results
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifical (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Tecnical faisability and financial support will be discussed before mandatory contractualization.